CLINICAL TRIAL: NCT00895024
Title: Caregiver Assessments of the Quality of Home Hospice Care: A Comparison Across 3 Ethnic Groups (A Preliminary Study)
Brief Title: Caregiver Assessments of the Quality of Home Hospice Care
Status: Terminated | Type: Observational
Why Stopped: PRMS No Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2009-0031
Record Dates: First submitted 2009-05-05; First posted 2009-05-07 (Estimated); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Advanced Cancer
Keywords: Caregiver; Questionnaire; Home Hospice Care; Family Evaluation of Hospice Care; FEHC; The Texas Revised Inventory of Grief; TRIG; Cross-ethnic differences; Parenteral Hydration; Grief
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Caregivers
  Interventions: Behavioral: Phone Interview/Questionnaire

INTERVENTIONS:
Behavioral: Phone Interview/Questionnaire — 35-minute questionnaire over the phone.
  Other Names: Survey

SUMMARY:
The Objectives are to administer the Family Evaluation of Hospice Care (FEHC) questionnaire and The Texas Revised Inventory of Grief (TRIG) to caregivers previously enrolled into the parent grant and conduct supplemental analyses to:

1. examine cross-ethnic differences in the caregivers' quality of hospice care assessments.
2. investigate the association between parenteral hydration status of the patient and the quality of care assessments provided by the caregivers after death.
3. examine the association between levels of grief (as measured by the TRIG) and the quality of hospice care assessments provided by the caregiver.

DETAILED DESCRIPTION:
After the death of their loved-ones, caregivers will be asked to report on the care received by their care recipient and the quality of practical and emotional care provided to them by hospice by completing the 25-minute FEHC questionnaire over the phone. Caregivers will also be asked 16 additional questions to assess their attitudes and beliefs about hydration at the end of life, and a brief questionnaire to assess past and current levels of grief (TRIG). The additional questions on hydration and grief can easily be completed in less than 10 minutes over the phone. The entire interview should take no more than 35 minutes to complete.

Bereaved caregivers who have participated in the parent grant and have lost their loved one within 3-23 months will be mailed a letter from Drs. Bruera and Torres inviting them to participate in the voluntary supplemental after-death survey. The letter will include a brief description of the research study and appropriate contact information for the caregiver to call if she/he is interested in participating. The letters then will be followed up by a phone call from Dr. Torres to verify receipt of the letter. If the caregivers express their interest in participating in the study, they will be asked a few screening questions over the phone to verify their eligibility. Once found eligible for the study, a telephone verbal consent will be obtained.

Dr. Isabel Torres will conduct the phone interviews with 128 primary caregivers who had previously completed the parent grant protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Bereaved family caregivers who completed their participation in the parent protocol (2006-0494) and have lost their loved one within 3-23 months.
2. Caregivers who participated in the parent grant met the inclusion/exclusion criteria of the parent grant.

Exclusion Criteria:

1. Bereaved family caregivers who did not complete their participation in the parent protocol or any other caregiver who was never enrolled in the parent protocol (2006-0494).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Bereaved family caregivers who completed their participation in the UT MDACC parent protocol (2006-0494) and have lost their loved one within 3-23 months. Caregivers who participated in the parent grant met the inclusion/exclusion criteria of the parent grant.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
Survey assessment of cross-ethnic differences in caregivers' quality of hospice care | 3-23 Months After Hospice Care

CONTACTS AND LOCATIONS:
Overall Officials: Lorna H. McNeill, MPH, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org